CLINICAL TRIAL: NCT06565507
Title: A Double-blind Multicenter, Randomized Controlled Trial of Single and Multiple Dose Regimens of Oxfendazole for Mild (One or Two Lesions) Parenchymal Brain Cysticercosis, With an Open Comparison Group
Brief Title: Oxfendazole in Mild Parenchymal Brain Cysticercosis
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universidad Peruana Cayetano Heredia (Other)
Collaborators: Oxfendazole Development Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 211661
Record Dates: First submitted 2024-08-12; First posted 2024-08-22 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-06

CONDITIONS: Brain Cysticercosis
Keywords: Cysticercosis; Cysticercosis treatment
MeSH Terms: conditions — Neurocysticercosis; Cysticercosis | interventions — oxfendazole; Albendazole

STUDY DESIGN:
Intervention Model Description: The intervention administered orally will be done randomly, in three groups or arms; arms 1 and 2, receiving oxfendazole (OXF) in a single dose or oxfendazole in three-days regimen (days 1, 4 and 7), respectively; arm 3, receiving a ten days albendazole (ABZ) + praziquantel (PZQ) regimen.
Who Masked: Participant, Investigator
Masking Description: This study is a double-blind trial in regards to dose regime of OXF. Neither the investigators nor the subjects know which dose of OXF a given subject is receiving, although subjects and clinical study staff will know whether they are receiving one of the OXF regimes or active ABZ+PZQ.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Intervention 1 (Experimental): OXF 20 mg/kg/d, single dose, orally
  Interventions: Drug: Oxfendazole single dose
- Intervention 2 (Experimental): OXF 20 mg/kg/d, for three days (1, 4 and 7), orally
  Interventions: Drug: Oxfendazole three doses
- Comparison regimen (Active Comparator): Combined treatment with albendazole (15 mg/k/d) plus praziquantel (50 mg/k/d), for 10 days, orally.
  Interventions: Drug: albendazole plus praziquantel regime

INTERVENTIONS:
Drug: Oxfendazole single dose — Subjects will receive active oxfendazole, 20 mg/kg/day, orally, as a single dose. Oxfendazole placebo will be used at days 4 and 7 to maintain blinding between the two intervention arms.
  Other Names: Intervention 1
  Arms: Intervention 1
Drug: Oxfendazole three doses — Subjects will receive active oxfendazole, 20 mg/kg/day, orally, in three days (1, 4 and 7)
  Other Names: Intervention 2
  Arms: Intervention 2
Drug: albendazole plus praziquantel regime — Subjects will receive a combination of albendazole plus praziquantel, as a standard treatment for brain cysticercosis (neurocysticercosis), orally, for ten days. Albendazole will be given at 15/kg/d and praziquantel at 50/kg/d.
  Other Names: Comparison regimen
  Arms: Comparison regimen

SUMMARY:
The goal of this clinical trial is to compare a single and multiple dose regimens of oxfendazole with the standard treatment in patients with mild (one or two lesions) parenchymal brain cisticercosis. The main question it aims to answer is if OXF will enhance clearance of brain parasites and therefore provide greater cysticidal efficacy, with the potential to provide a single-dose therapy for this type of NCC.

The study cohort will also allow us to identify early imaging markers that predict lesion resolution, as well as factors associated with residual calcification or focal gliosis after lesion resolution. This study will also provide additional information on the safety of the study interventions.

DETAILED DESCRIPTION:
This three-arm randomized controlled phase II/III clinical trial will compare the efficacy and safety of a single-dose regimen with 20 mg/kg oxfendazole and a regimen with three similar doses spread over seven days (day 1, day 4 and day 7), with the most effective antiparasitic regimen available, combined albendazole plus praziquantel for ten days in individuals with mild NCC (with one to two lesions).

Participants will receive treatment with oxfendazole (one or three dose regimens) or the standard treatment (albendazole + praziquantel). At day 15 after treatment onset, an MRI will be perfomed to evaluate early predictors of lesion resolution. MRI at day 90 will serve to evaluate efficacy (lesion resolution) and a day 180 MRI will evaluate sequelar lesions. CT will be perfomed at the en of the study to confirm persistence of calcified sequelar lesion.

The study will enroll 544 patients with viable or degenerating parenchymal NCC with no more than two lesions, all in a single brain area. Lesions can be one or two adjacent, viable or degenerating NCC lesions. Patients with only calcified lesions will not be included even if they show perilesional contrast enhancement.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female individuals between 12 and 75 years of age, with suspected viable or degenerating intraparenchymal brain cysticercosis on neuroimaging (CT or MRI) and fulfill the diagnostic criteria for solitary cysticercus granuloma (Rajshekhar and Chandy, 1997)
2. If female of child-bearing potential and men, willing to use an adequate method of contraception*, including implants, injectables, combined oral contraceptives, effective intrauterine devices, sexual abstinence, or vasectomized partner while participating in the study.
3. Patients with normal laboratory values for hemoglobin, platelet counts, total white blood cells, glucose, creatinine, bilirubin, ALT, and AST.
4. Availability to grant informed consent if you are over 18 years of age or assent if you are a minor between 12 and 17 years of age.

Exclusion Criteria:

1. Multiple lesion sites or more than two adjacent lesions.
2. Suspected neurotuberculosis (Rajshekhar's criteria) [66,67]
3. More than two viable brain cysts.
4. Large brain cysts (> 3cm in diameter)
5. Subarachnoid neurocysticercosis or intraventricular
6. Untreated ocular cysticercosis
7. Previous therapy with ABZ (does not include patients who received single-dose 400 mg ABZ for intestinal parasites), or PZQ in the past twelve months.
8. Active pulmonary tuberculosis evidenced by a positive chest X-ray and positive sputum smears.
9. Systemic disease other than NCC that may affect therapy or short-term prognosis, including but not limited to chronic renal failure, hepatic insufficiency, cardiac failure, and steroid-dependent immune diseases.
10. Patients in unstable condition or with severe intracranial hypertension (ICH). Definition of severe ICH for this study would be the presence of headaches, nausea, and vomiting, and papilledema at fundoscopic examination.
11. Pregnancy
12. History of hypersensitivity to ABZ or PZQ
13. Concurrent treatment with cimetidine, ranitidine, or theophylline.
14. Chronic alcohol or drug abuse
15. Positive to Strongyloides infection
16. History of reported allergy to contrast substances used in MRI.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 544 (Estimated)
Dates: Start 2024-12-15 (Estimated); Primary Completion 2028-03-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy: completely resolution or persistance only as small lesion remnants. | Three months after treatment onset
  Proportion of participants whose lesions completely resolved or persist only as small lesion remnants (<20% of the original lesion size).

SECONDARY OUTCOMES:
Clinical effectiveness: Seizure relapses. | In the initial 12 months after treatment
  The frequency of seizure relapses in individuals whose lesions resolved compared to those who had remaining viable or degenerating lesions on month 3 MRI
Safety: Serious adverse events | In the initial 12 months after treatment
  Proportion of participants in each group who develop serious or severe adverse events, and the numbers of adverse events per group

OTHER OUTCOMES:
Early imaging markers predicting lesion resolution. | Month 3
  Imaging characteristics on MRI at day 15 after treatment onset that are associated with successful lesion resolution on MRI.
Antiparasitic treatment type associated with gliosis or residual calcification. | Month 6 and month 12
  Antiparasitic treatment type (oxfendazole single dose, or oxfendazole three doses, or combined albendazol plus praziquantel treatment) associated with focal gliosis or residual calcification.
Antiparasitic treatment type associated with seizure relapses. | During the initial 12 months after antiparasitic treatment.
  Antiparasitic treatment type (oxfendazole single dose, or oxfendazole three doses, or combined albendazol plus praziquantel treatment) associated with seizure relapses.
Quality of life in Epilepsy (QOLIE-31) score around antiparasitic treatment in NCC, to assess emotional and psychological effects, and medical and social effects. | Before treatment and 12 months after antiparasitic treatment.
  Factors associated with reduced quality of life before and after anti-parasitic treatment for mild parenchymal NCC
Cysticercus size associated with seizure relapses. | During the initial 12 months after antiparasitic treatment.
  Measururement of cysticercus size, in millimeters, to evaluate its association with seizure relapses.
Number of baseline seizures associated with seizure relapses. | During the initial 12 months after antiparasitic treatment.
  Number of pre-treatment seizures associated with seizure relapses after initiation of antiparasitic treatment.
Cysticercus size associated with gliosis or residual calcification. | Month 6 and month 12
  Measururement of cysticercus size, in millimeters, to evaluate its association with gliosis or residual calcification.

CONTACTS AND LOCATIONS:
Overall Officials: Hector H Garcia, MD, PhD, Principal Investigator — Universidad Peruana Cayetano Heredia